CLINICAL TRIAL: NCT00122603
Title: Efficacy and Safety of Regimens Restricted to a Combination of Two Boosted Protease Inhibitors as Potent Antiretroviral Therapy in HIV-1 Infected Patients. ANRS 127 2IP
Brief Title: Dual Boosted Protease Inhibitor Regimens Without Any Additional Antiretroviral Therapy in HIV-1 Infected Patients (ANRS127)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Bristol-Myers Squibb (Industry); GlaxoSmithKline (Industry); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-003470-20; ANRS 127 2 IP
Record Dates: First submitted 2005-07-19; First posted 2005-07-22 (Estimated); Last update posted 2011-12-22 (Estimated); Status verified 2011-12

CONDITIONS: HIV Infections
Keywords: HIV Protease Inhibitors; HIV infections; Atazanavir; Saquinavir; Fosamprenavir; ritonavir; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — fosamprenavir; Saquinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Atazanavir + Fosamprenavir + ritonavir
  Interventions: Drug: Fosamprenavir
- group 2 (Experimental): Atazanavir + saquinavir + ritonavir
  Interventions: Drug: Saquinavir

INTERVENTIONS:
Drug: Fosamprenavir — ATV (150mg: 2 pills per day) + RTV (100mg: 1 pill twice a day) + FPV (700mg: 1 pill twice a day)
  Arms: Group 1
Drug: Saquinavir — ATV (150mg: 2 pills per day) + RTV (100mg: 1 pill per day) + SQV (500mg: 3 pills per day)
  Arms: group 2

SUMMARY:
The purpose of this study is to evaluate virological efficacy and safety of two double protease inhibitor regimens: atazanavir/fosamprenavir/ritonavir 300 mg once daily/ 700/100 mg twice daily, versus atazanavir/saquinavir/ritonavir 300/1500/100 mg once daily in protease inhibitor naive HIV-1 patients.

DETAILED DESCRIPTION:
The purpose of this randomized, open-label study is to evaluate virological efficacy and safety of two double protease inhibitor regimens: atazanavir/fosamprenavir/ritonavir 300 mg once daily/ 700/100 mg twice daily, versus atazanavir/saquinavir/ritonavir 300/1500/100 mg once daily in protease inhibitor naive HIV-1 patients.

Patients with CD4 cell counts over or equal to 200/mm3, HIV viral load between 10,000 and 750,000 copies per milliliter, and wild-type genotype at baseline will be eligible. This multicenter study will enroll 60 patients (n=30 in each group). The planned duration of the study is 48 weeks from the enrolment of the last subject.

The primary efficacy endpoint will be virologic success defined as HIV RNA levels below 50 copies/ml after 16 weeks of initial treatment. The durability of this response will be evaluated and patients will be followed for 48 weeks.

The primary safety endpoint will be treatment interruptions because of adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Protease inhibitor naive patients
* Wild type genotype
* CD4 greater than 200/mm3
* Viral load between 10,000 copies/ml and 750,000 copies/ml
* Signed informed consent

Exclusion Criteria:

* Pregnancy; breast feeding
* Antiretroviral (ARV) pretreated patients
* Hyperlipidemic treatment
* Evolutive disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2005-12; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Virologic success defined as HIV RNA levels below 50 copies/ml after 16 weeks of initial treatment

SECONDARY OUTCOMES:
Safety of protease inhibitors
Percentage of patients with viral load below 400 copies/ml at week 16 (W16)
Body mass index (BMI)

CONTACTS AND LOCATIONS:
Overall Officials: Roland Landman, MD, Principal Investigator — Hopital Bichat SMIT A Paris; Jean Pierre Aboulker, MD, Study Chair — Inserm SC10
Locations (1):
- Service des Maladies infectieuses et tropicales Hopital Bichat Claude Bernard, Paris, France

REFERENCES:
- [Derived] Landman R, Capitant C, Descamps D, Chazallon C, Peytavin G, Katlama C, Pialoux G, Bentata M, Brun-Vezinet F, Aboulker JP, Yeni P; ANRS 127 Study Group. Efficacy and safety of ritonavir-boosted dual protease inhibitor therapy in antiretroviral-naive HIV-1-infected patients: the 2IP ANRS 127 study. J Antimicrob Chemother. 2009 Jul;64(1):118-25. doi: 10.1093/jac/dkp146. Epub 2009 May 6. PMID 19420019